CLINICAL TRIAL: NCT02881437
Title: Assessment of the IgG Trough Level in Subjects With Primary Immunodeficiency Switching From Standard Subcutaneous Immunoglobulin (SCIG) to Every Other Week HyQvia
Brief Title: IgG Level in Primary Immunodeficiency Switching From Standard SCIG to Every Other Week HyQvia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015_31; 2016-001480-36 (EudraCT Number)
Record Dates: First submitted 2016-08-17; First posted 2016-08-29 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Primary Immunodeficiency
Keywords: Primary Immunodeficiency; SubCutaneous Immunoglobulins
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IgHy10 (HyQvia) (Experimental): Open-label, one arm study conducted in France in subjects with PI to IgG trough level at steady state after standard SCIG dosing and after IgHy10 (HyQvia) administered every other week and every 3-4 weeks at equivalent dose. The study will have three periods:
  * The first period is a one-week ramp-up period. The first administration of IgHy10 (HyQvia) will be with a one-week dose
  * During the first three-month follow-up period, IgHy10 (HyQvia) will be administered, every other week at a dose equivalent to the dose administered with the previous treatment (standard SCIG).
  * At the end of this first follow-up period, the dose of IgHy10 (HyQvia) will be increased for the next infusion to reach a 3-4 week equivalent dose.
  Interventions: Drug: IgHy10

INTERVENTIONS:
Drug: IgHy10 — Sub Cutaneous IgHy10 administration
  Other Names: HyQvia

SUMMARY:
Most immunodeficiencies are related to severe immunoglobulin deficiencies which require lifelong replacement therapy with immunoglobulin G (IgG) to reduce the incidence and severity of infections. IgG can be administered intravenously (IGIV) every 21 or 28 days or subcutaneously every week or every other week (IGSC) for subjects who do not tolerate IV infusions or have difficulties with venous access. No head-to-head data are available to directly compare HyQvia with conventional SCIG. However, SCIG is indicated for administration frequencies from daily up to every other week dosing while HyQvia is indicated for infusion frequencies every 2-4 weeks. This study is designed to assess the IgG trough level after switching from standard SCIG to every other week HyQvia and HyQvia every 3-4 weeks

DETAILED DESCRIPTION:
Open-label, one arm study conducted in France in subjects with PI to IgG trough level at steady state after standard SCIG dosing and after HyQvia administered every other week and every 3-4 weeks at equivalent dose. The study will have three periods:

* The first period is a one-week ramp-up period. The first administration of HyQvia will be with a one-week dose as specified in the summary of product characteristics of HyQvia.
* During the first three-month follow-up period, HyQvia will be administered, every other week at a dose equivalent to the dose administered with the previous treatment (standard SCIG).
* At the end of this first follow-up period, the dose of HyQvia will be increased for the next infusion to reach a 3-week equivalent dose. If it this volume is well tolerated, the following dosing will be a 4-week equivalent dose. HyQvia will then be administered every 3 or 4 weeks for three months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years old at the time inclusion.
* Suffering from PI requiring immunoglobulin replacement therapy.
* Treated with SCIG at stable dose for at least 3 months at the time of inclusion.
* Well balanced SCIG treatment according to the investigator at the time of inclusion.
* If female of childbearing potential, the subject must have a negative blood or urine pregnancy test at the time of inclusion and must agree to employ adequate birth control measures during the whole study.
* Willing and able to comply with the requirements of the protocol.
* Having signed the informed consent form.

Exclusion Criteria:

* Known history of chronic kidney disease, or glomerular filtration rate (GFR) of <60 mL/min/1.73m2 estimated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at the time of screening.
* Having received a chemotherapy or immunomodulating therapy for either malignant or chronic inflammatory disease for over 6 months.
* Receiving anticoagulant therapy.
* Having abnormal protein loss (protein losing enteropathy, nephrotic syndrome).
* Know allergy to hyaluronidase.
* Family member or employee of the investigator.
* Having participated in another interventional clinical study involving an investigational product (IP) or investigational device within 30 days prior to inclusion or scheduled to participate in another clinical study involving an another investigational product or investigational device during the course of this study.
* If female, pregnant or breastfeeding at the time of enrolment.
* If female, planning to become pregnant during the time period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in IgG trough level at 3 months (visit 3) as compared to baseline (visit 1). | Every 2 weeks during the baseline (visit 1) and the 3 months (visit3)

SECONDARY OUTCOMES:
The change in IgG trough level at 6 months (visit 4) as compared to baseline (visit 1) and 3 months (visit 3). | Every 3 weeks after the 3 months (visit 3) as 6 months ( visit 4)
Number of adverse reactions | 6 months
Incidence rate of adverse reactions | 6 months
Number of infection | 6 months
The Short Form (36) Health Survey | at 6 months
  standardized test for measuring the quality of life
Treatment Satisfaction Questionnaire for Medication (TSQM-9). | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hachulla, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - CHRU, Hôpital Claude Huriez, Lille
  - Hôpital de la Conception, Marseille
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital St Louis, Paris
  - Hôpital Necker, Paris
  - Hôpital Haut Lévèque, Pessac
  - CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No